CLINICAL TRIAL: NCT04957147
Title: The REMIT-DCM Study: Reverse Remodelling and Remission Markers in the Serial Evaluation of Recent-onset Dilated Cardiomyopathy
Brief Title: Reverse Remodelling and Remission Markers in the Serial Evaluation of Recent-onset Dilated Cardiomyopathy
Acronym: REMIT-DCM
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19IC5198
Record Dates: First submitted 2021-06-22; First posted 2021-07-12 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Dilated Cardiomyopathy
Keywords: Dilated cardiomyopathy; Left ventricular reverse remodelling; Heart failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: patients with dilated cardiomyopathy: Patients with recent-onset dilated cardiomyopathy
  Interventions: Other: 12 months of guideline-directed heart failure therapy
- Group B: healthy volunteers: Healthy volunteers with no known heart disease

INTERVENTIONS:
Other: 12 months of guideline-directed heart failure therapy — Standard guideline-directed heart failure drug +/- device therapy
  Groups: Group A: patients with dilated cardiomyopathy

SUMMARY:
Approximately 30-40% of patients with non-ischaemic dilated cardiomyopathy (DCM) undergo significant left ventricular reverse remodelling in response to guideline-directed therapies. This is characterised by improvement in systolic dysfunction and regression of left ventricular dilatation. In some patients, extensive left ventricular reverse remodelling is accompanied by resolution of symptoms and normalisation of cardiac biomarkers, resulting in a state of clinical remission.

The mechanistic drivers behind left ventricular reverse remodelling and clinical remission are poorly understood. Current techniques to predict ventricular remodelling trajectory and clinical remission in patients with recent-onset DCM are limited.

The purpose of this study is to characterise predictors and markers of left ventricular reverse remodelling and clinical remission in patients with recent-onset DCM using molecular markers, genetics and advanced CMR imaging.

DETAILED DESCRIPTION:
The REMIT-DCM study is a single-centre pilot observational cohort study. 70 patients with recent-onset DCM (Group A) and up to 40 healthy volunteers (Group B) will be recruited. Patients with DCM will be recruited over a 2-year period and will be followed up for 12 months. Subjects in Group A may be offered an optional further study visit at 24-48 months after enrolment in order to assess whether cardiac remodelling and clinical remission are sustained over the intermediate-term.

Patients with DCM (Group A) will attend 3 study visits at The Royal Brompton Hospital (baseline, 2-3 months and 12 months). Each study visit will involve a clinical consultation, blood sample collection (including routine clinical blood tests and sample storage for exploratory biomarkers), urine sample collection, 12-lead ECG, health questionnaire completion and a cardiovascular magnetic resonance scan (CMR). If patients are unable to have a CMR, 3D transthoracic echocardiography will be performed.

Healthy volunteers will attend a single study visit at The Royal Brompton Hospital. This will involve a clinical consultation, blood sample collection (including routine clinical blood tests and sample storage for exploratory biomarkers), urine sample collection, 12-lead ECG, health questionnaire completion and a CMR.

ELIGIBILITY:
For DCM cohort (Group A):

Inclusion Criteria:

* Age ≥16.
* Able to give informed consent.
* Confirmed DCM with symptom-onset within the last 6 months and LVEF ≤ 45%. The diagnosis of DCM will be confirmed using the European Society of Cardiology definition, based on reduced LVEF and elevated LV end-diastolic volume indexed to body surface area, compared to published age- and sex-specific reference values

Exclusion Criteria:

* Significant coronary artery heart disease, defined as a stenosis of >50% of an epicardial coronary artery affecting the proximal or mid-portion of the vessel on invasive angiography or computed tomography coronary angiography (CTCA), previous percutaneous coronary intervention, CMR late gadolinium enhancement pattern suggestive of previous myocardial infarction of ≥ 2 segments of ≥ 50% transmural infarction of the LV wall.
* High suspicion of concomitant hypertrophic cardiomyopathy, amyloidosis, Fabry disease, sarcoidosis, active myocarditis, Chagas disease or hemochromatosis.
* History of primary valvular heart disease or congenital heart disease.
* Severe, untreated or untreatable hypertension (systolic blood pressures routinely >180 mm Hg and/or diastolic blood pressures >120 mm Hg)
* Pregnancy and/or breastfeeding.
* Severe renal disease (GFR <15 mls/min).

For healthy volunteer cohort (Group B):

Inclusion Criteria:

* Age ≥16.
* Able to give informed consent.

Exclusion criteria:

* Participants with any clinically significant cardiovascular or metabolic disease.
* Participants taking prescription medicines for significant cardiovascular or metabolic disease.
* Female subjects if they are pregnant or breastfeeding at the time of recruitment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group A: There are 3 routes via which patients with DCM may be recruited:
  1. Patients from the Royal Brompton & Harefield NHS Trust clinical service (inpatients, patients from clinics and patients referred for a CMR).
  2. Patients with DCM may also be recruited from collaborating district general hospitals, defined as Patient Identification Centres (PICs). Clinicians at these sites have agreed to identify suitable patients encountered within their routine practice.
  3. Patients will be able to self-refer via The Heart Hive for consideration by the study team. The Heart Hive (https://www.thehearthive.org/) is an online platform that offers patients with cardiomyopathy and healthy volunteers the opportunity to connect with researchers regarding participation in research studies.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical remission | 12-months
  If all 3 of the following criteria are met at 12-month assessment:
  i. Increase in left ventricular ejection fraction (LVEF) by ≥ 10% to a value ≥ 50% and decrease in indexed left ventricular end diastolic volume (LVEDV) to within normal range according to age-/sex-corrected normograms.
  ii. NYHA class I.
  iii. NT-Pro BNP <250 ng/L.

SECONDARY OUTCOMES:
Left ventricular reverse remodelling | 12-months
  Evaluated by changes in indexed left ventricular end systolic volume (LVESV), indexed LVEDV and LVEF between baseline and 12 months.
Left ventricular reverse remodelling | 12-months
  Evaluated using a pre-specified threshold: patients with DCM will be divided into 2 groups at the 12-month timepoint:
  i. Left ventricular reverse remodelling: an increase in LVEF by ≥ 10% to a value ≥ 40%; and a decrease in indexed LVEDV by ≥ 10%.
  ii. No left ventricular reverse remodelling: no increase in LVEF by ≥ 10% to a value ≥ 40% and/or no decrease in indexed LVEDV by ≥ 10%.
Major adverse cardiovascular events | 12-months
  Composite of cardiovascular death, major heart failure or major arrhythmic events.
Change in health status using Kansas City Cardiomyopathy questionnaire | 12-months
  Change in Kansas City Cardiomyopathy questionnaire scores from baseline to 12-months
Change in health status using SF-12 questionnaire | 12-months
  Change in SF-12 questionnaire scores from baseline to 12-months
Change in health status using EQ-5D questionnaire | 12-months
  Change in EQ-5D questionnaire scores from baseline to 12-months
Sustained clinical remission at 24-48 months after enrolment | 48 months
  For those in clinical remission at 12-month timepoint, the proportion that have sustained clinical remission at 24-48 months after enrolment.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay K Prasad, Principal Investigator — Imperial College London
Locations (1):
- Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No